CLINICAL TRIAL: NCT06972589
Title: The Effect of Mask Design on Ventilation Parameters in COPD and OHS Patients on Long-term Home Non-invasive Ventilation. An Experimental Study.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: U1111-1322-0270; CIA-356 (Other: Fisher and Paykel Healthcare)
Record Dates: First submitted 2025-05-07; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease); Obesity Hypoventilation Syndrome (OHS)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Obesity Hypoventilation Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Noninvasive ventilation (CPAP or bilevel) with the investigational mask (Experimental)
  Interventions: Device: Investigational Mask
- Noninvasive ventilation (CPAP or bilevel) with the conventional mask (Active Comparator)
  Interventions: Device: Conventional mask

INTERVENTIONS:
Device: Investigational Mask — Wear mask to enable the delivery of noninvasive ventilation (CPAP or bilevel) therapy during sleep.
  Arms: Noninvasive ventilation (CPAP or bilevel) with the investigational mask
Device: Conventional mask — Wear mask to enable the delivery of noninvasive ventilation (CPAP or bilevel) therapy during sleep.
  Arms: Noninvasive ventilation (CPAP or bilevel) with the conventional mask

SUMMARY:
Chronic obstructive pulmonary disease (COPD) and obesity hypoventilation syndrome (OHS) are respiratory conditions that disrupt normal breathing. Positive airway pressure, specifically Non-Invasive Ventilation (NIV) delivers positive pressures via an interface such as a face mask and has been shown to improve breathing and reduce symptoms in patients with these conditions. Regular use of NIV can lead to better symptom management, improved quality of life, and reduced use of healthcare resources. However, poor performance of the NIV mask and poor comfort can make NIV therapy harder to tolerate. This study will assess if a new mask helps to improve the breathing of people on NIV and normalize blood gases.

DETAILED DESCRIPTION:
Participants are moved to the sleep laboratory for the night where they are provided with beds.

* The participants are put on their prescribed airway pressure support with the first randomized mask.
* After at least 60 minutes of recording, participants are awakened to switch back to the second mask. They are then allowed to sleep uninterrupted for the rest of the night.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Prescribed nocturnal NIV for COPD or OHS
* Able to complete an overnight sleep study
* Comfortable to sleep on a standard double bed
* Capacity to complete informed consent

Exclusion Criteria:

* Uncontrolled sleep apnea (Apnea-hypopnea index (AHI) over 15 events/hour off personal NIV device data)
* Prescribed IPAP above 25 cmH2O
* Allergic to adhesive of the sensors
* Self-reported cold/flu symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in respiratory rate | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: William Good, Medical degree, Principal Investigator — Middlemore Hospital, New Zealand
Locations (1):
- Fisher and Paykel Healthcare Sleep Laboratory, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No